CLINICAL TRIAL: NCT06487455
Title: An Open, Multicenter, Dose-escalation, and Dose-expansion Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Initial Efficacy of SPH7485 Tablets in Patients With Advanced Solid Tumors.
Brief Title: A Clinical Study of SPH7485 Tablets in the Treatment of Advanced Solid Tumors.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Pharmaceuticals Holding Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPH7485-101
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SPH7485 (Experimental)
  Interventions: Drug: SPH7485

INTERVENTIONS:
Drug: SPH7485 — SPH7485： Orally, once daily, 50-400mg, 21 days per cycle

SUMMARY:
To evaluate the efficacy and safety of SPH7485 tablets in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed advanced solid tumors；
2. At least one extracranial measurable lesion;
3. ECOG (Eastern Cooperative Oncology Group) performance status score of 0 or 1;
4. Subjects whose laboratory examination indicators meet the prescribed standards during the screening period;
5. Life expectancy≥3 months;
6. Subjects whose toxic reactions to previous antitumor therapy returned to baseline or CTCAE≤grade 1;
7. Female subjects whose pregnancy tests are negative; Male subjects agree not to donate sperm; Subject and partner agree to use reliable contraception;
8. Volunteer to participate in clinical research; Fully understand and know the study and sign the informed consent; Subjects willing to follow and able to complete all test procedures.

Exclusion Criteria:

1. Subjects who have received the prescribed other anti-tumor treatments at the prescribed time prior to the first dose;
2. Subjects who have received previous drugs with the same target;
3. Subjects with active infections requiring systemic treatment;
4. Subjects with third gap fluid accumulation that cannot be controlled by drainage or other methods;
5. Subjects with uncontrolled or severe cardiovascular disease;
6. Severe lung disease;
7. Subjects with conditions that may affect the absorption, distribution, metabolism, or excretion of the test drug;
8. Subjects taking strong/moderate inhibitors or inducers of CYP3A4;
9. Subjects who use or require long-term use of hormonotherapy before screening;
10. Subjects who have had other malignancies within the past 5 years;
11. Subjects with symptomatic CNS metastasis, pial metastasis, or spinal cord compression due to metastasis;
12. Subjects who have undergone or are scheduled to undergo major surgery, or have not yet recovered from surgery;
13. Abnormal virological examination during screening; History of immune deficiency;
14. Uncontrolled systemic diseases;
15. Subjects who have participated in any other clinical trial and received treatment within 21 days prior to the first dose;
16. Subjects who have received or plan to receive live or attenuated vaccines within 28 days prior to first dose;
17. Subjects with a history of severe allergy or known allergy to this product and its excipients;
18. Subjects who cannot follow the study protocol to complete the required study visit and dosing;
19. Subjects with a history of alcohol or drug abuse;
20. Lactating female patients;
21. Subjects with a clear past history of neurological or psychiatric disorders. Subjects with primary diseases of other vital organs deemed unsuitable for inclusion by the investigator;
22. Subjects deemed unsuitable for this clinical study by the investigator for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2024-08-06 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
DLT(Dose-limiting toxicity) | Approximately 24 days
  Measurement of DLT of SPH7485 in all subjects
Maximum tolerated dose（MTD） | Approximately 24 days
  Measurement of MTD of SPH7485 in all subjects
Incidence of Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Approximately 2 years
  Incidence of Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)

SECONDARY OUTCOMES:
ORR(Objective Response Rate) | Approximately 2 years
  Tumor response will be evaluated according to the Response Evaluation Criteria Solid Tumors (RECIST) criteria version 1.1.
DoR(Duration of response) | Approximately 2 years
  DOR was defined as the time interval between the date of the first documented response (CR or PR) and the date of the first documented disease progression or death due to any cause
DCR(Disease Control Rate) | Approximately 2 years
  DCR was defined as the percentage of patients who have achieved complete response, partial response and stable disease
PFS(Progression-free survival) | Approximately 2 years
  PFS was defined as the time interval between study treatment initiation and the first occurrence of progression disease or death, whichever occurred first.
PK(Pharmacokinetics):Tmax | Approximately 3 days
  Time to peak plasma concentration (Tmax)
PK(Pharmacokinetics):Cmax | Approximately 3 days
  Maximum serum concentration(Cmax)
PK(Pharmacokinetics):AUC | Approximately 3 days
  Area under the plasma concentration versus time curve (AUC)

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - XiangYa Hospital CentralSouth University, Changsha
  - Fujian Cancer Hospital, Fuzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Yunnan Cancer Hospital, Kunming
  - Fudan University Shanghai Cancer Center, Shanghai
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan